CLINICAL TRIAL: NCT04515680
Title: National Survey on Endocrine Function and Bone Metabolism in Transfusion--dependent Patients Treated With Deferasirox
Brief Title: Endocrine Function During Deferasirox Therapy
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Silverio Perrotta, Prof., University of Campania Luigi Vanvitelli
Other Study IDs: CICL670AIT16T
Record Dates: First submitted 2020-08-06; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Iron Overload; Transfusion-dependent Thalassemia; Endocrine; Complications
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A national survey on the prevalence and natural history of endocrine complications in thalassemia transfusion--dependent patients treated with deferasirox was designed, in order to assess a larger population during a longer follow up and improve the quality of previous investigations.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric patients with transfusion---dependent thalassemia;
* Chelation with deferasirox as assigned chelation therapy;
* Available medical history including relevant clinical data (age at start of transfusion regimen, age at start of chelation therapy, prior chelation therapy, concomitant diseases and concomitant treatments, including hormonal replacement treatments if appropriate) and laboratory data (e.g TSH, FT3 and FT4, fasting serum glucose, OGTT serum glucose, bone mineral density z---score, T---score, g/cm2, PTH, FSH, LH, testosterone and estradiol, serum ferritin, liver function tests,renal function tests, MRI T2* value) at baseline and at the end of study

Exclusion Criteria:

* Non transfusion- dependent patients;
* Other chelation therapy than deferasirox or combination with other chelators during the observation;
* Absence of complete medical history as above specified

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients visited at the participating sites since September 2009 were recruited into the cohort provided the inclusion criteria were met: affected by TDT and on deferasirox monotherapy during the study period.
Sampling Method: Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline number of endocrine disorders at study completion | baseline through study completion, a minimum of 5 years
  Absolute change in number of patients diagnosed with any endocrine disorder at the baseline and at the study completion

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi della Campania Luigi Vanvitelli, Naples, Italy